CLINICAL TRIAL: NCT02241785
Title: A Phase 4 Multicenter, Open-Label, Single Arm Study to Evaluate Switching From BRACET/Gilenya® to Natalizumab in Subjects With Relapsing Forms of Multiple Sclerosis (MS)
Brief Title: Natalizumab as an Efficacy Switch in Participants With Relapsing Multiple Sclerosis After Failure on Other Therapies
Acronym: ESCALATE
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Business Decision
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 101MS409; 2013-005586-39 (EudraCT Number)
Record Dates: First submitted 2014-09-12; First posted 2014-09-16 (Estimated); Results first posted 2017-06-05 (Actual); Last update posted 2017-06-05 (Actual); Status verified 2017-04

CONDITIONS: Relapsing Multiple Sclerosis
MeSH Terms: interventions — Natalizumab

ARMS (1):
- natalizumab (Experimental): natalizumab 300 mg intravenously (IV) every 4 weeks
  Interventions: Drug: natalizumab

INTERVENTIONS:
Drug: natalizumab — Administered as specified in the treatment arm
  Other Names: BG00002; Tysabri

SUMMARY:
The primary objective of the study is to determine the efficacy of natalizumab (Tysabri, BG00002) in participants with relapsing forms of multiple sclerosis (MS) who have failed Gilenya or BRACET (Betaseron, Rebif, Avonex, Copaxone, Extavia, Tecfidera) as measured by the proportion of participants with no evidence of disease activity (NEDA) at Year 1. The secondary objectives in this study population are: change in total T1 hypointense and total T2 hyperintense lesion volume; proportion of participants with NEDA at Year 2; evaluation of the impact of natalizumab on annualized relapse rate (ARR); and change in Multiple Sclerosis Impact Scale-29 (MSIS-29) physical impact score.

ELIGIBILITY:
Key Inclusion Criteria:

* Subjects of childbearing potential must practice effective contraception from Day -1 and be willing and able to continue contraception for duration of the study.
* Must have documented diagnosis of relapsing MS (McDonald 2010 Criteria [Polman 2011]) at Screening.
* Must have been treated with Gilenya or Betaseron, Rebif, Avonex, Copaxone, Extavia, Tecfidera (BRACET) for at least the 12 months prior to Screening with no interruption of treatment greater than 1 month. Prior treatment with natalizumab is allowed; however, there must be a minimum 1 year since last natalizumab infusion and the Screening visit of this study, and if discontinuation of natalizumab in the past was not due to intolerance, anti-natalizumab antibodies, or efficacy loss.
* Must have had disease activity in the 6 months prior to Screening while on Gilenya or BRACET (as defined by at least 1 gadolinium enhancing lesion OR at least 2 new T2 lesions compared with magnetic resonance imaging done within 12 months of screening OR clinical relapse, or Expanded Disability Status Scale [EDSS] progression of 1 point)
* Must have an EDSS score from 0 to 5.5 inclusive at Screening.
* Must have lymphocyte count that is documented as at or above the lower limit of normal (LLN) by the day before the first Tysabri infusion. If lymphocytes have not returned to LLN or above the day before the first Tysabri infusion (day 0), the subject has screen failed. The subject who screen fails is eligible to undergo Rescreening once; if additional Rescreening is considered, please contact the study medical monitor.

Key Exclusion Criteria:

* History or positive test result at Screening for human immunodeficiency virus.
* History or positive test result at Screening for hepatitis C virus antibody or current hepatitis B infection (defined as positive for hepatitis B surface antigen and/or hepatitis core antibody).
* Prior treatment with natalizumab (either commercially or through a clinical study) within 1 year of Day -1.
* Contraindications to treatment with natalizumab as described in the Prescribing Information for each of the participating countries.
* Known allergy to natalizumab or any of its ingredients, or known to be anti-natalizumab antibody positive.
* Diagnosis of primary progressive MS, secondary progressive MS, and/or progressive-relapsing MS.
* An MS relapse that has occurred within the 30 days prior to Day -1 and/or the subject has not stabilized from a previous relapse prior to Day -1.
* Known active malignancies (subjects with cutaneous basal cell carcinoma that has been completely excised prior to study entry remain eligible).
* History of severe opportunistic infections (including progressive multifocal leukoencephalopathy) or any clinically significant cardiac, endocrinologic, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, and renal, or other major disease, as determined by the Investigator
* Clinically severe active infection within 1 month prior to Screening.
* Females breastfeeding, pregnant, or planning to become pregnant; women who are not post-menopausal or surgically sterile who are unwilling to practice contraception; women who have a positive pregnancy test result at Day -1.
* Prior history of immunosuppressant use (e.g., mitoxantrone, azathioprine, methotrexate, cyclophosphamide, mycophenolate, cladribine, rituximab) in the last 12 months prior to Screening. Prior history of alemtuzumab use at any point in the past.

NOTE: Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2014-09-30 (Actual); Primary Completion 2016-05-02 (Actual); Study Completion 2016-05-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (11):
- United States (11):
  - Research Site, Fullerton, California
  - Research Site, Aurora, Colorado
  - Research Site, Des Moines, Iowa
  - Research Site, St Louis, Missouri
  - Research Site, Plainview, New York
  - Research Site, Raleigh, North Carolina
  - Research Site, Akron, Ohio
  - Research Site, Cleveland, Ohio
  - Research Site, Knoxville, Tennessee
  - Research Site, Round Rock, Texas
  - Research Site, Tacoma, Washington

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Natalizumab
Started | 47
Completed | 0
Not Completed | 47
Not completed — Sponsor Termination | 43
Not completed — Withdrawal by Subject | 1
Not completed — Lost to Follow-up | 2
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Groups:
- Natalizumab: natalizumab 300 mg IV every 4 weeks
Arm/Group | Natalizumab
Number analyzed (Participants) | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.9 (10.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34
  Male | 13

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants With No Evidence of Disease Activity (NEDA) From Reset Baseline (Week 8) to Week 56
Description: The proportion of participants with NEDA, defined as follows: no Expanded Disability Status Scale (EDSS) progression (12-week sustained); no relapses; no gadolinium enhancing (Gd+) lesions; no new or enlarging T2 hyperintense lesions over 48 weeks after resetting the Baseline at Week 8 to remove contribution of combined unique active (CUA) lesions that occurred prior to Week 8, when natalizumab was not yet active. The EDSS quantifies disability in 8 functional systems. The final EDSS score is an ordinal clinical rating scale ranging from 0 (normal neurologic examination) to 10 (death due to MS) in half-point increments.
Time Frame: Reset Baseline (Week 8) to Week 56
Population: The limited number of participants enrolled and the early termination of the study resulted in efficacy data not collected, and efficacy outcomes not analyzed, as per the pre-specified plan of analysis.
Arm/Group | Natalizumab
Number analyzed (Participants) | 0

2. Secondary Outcome: Change in T1 Unenhancing Lesion Volume and T2 Lesion Volume From Baseline (Day -1) to Reset Baseline (Week 8)
Description: As measured by magnetic resonance imaging.
Time Frame: Baseline (Day -1) to Reset Baseline (Week 8)
Population: Intent-to-treat population: participants who received at least 1 infusion of study treatment and had an assessment.
Measure: Mean (Standard Deviation); unit: cc
Arm/Group | Natalizumab
Number analyzed (Participants) | 43
cc
  Change in T1 Unenhancing Lesion Volume | 0.11 (0.65)
  Change in T2 Lesion Volume | 0.01 (1.76)

3. Secondary Outcome: Proportion of Participants With NEDA From Week 8 (Reset Baseline) to Week 104
Description: Proportion of participants with NEDA from Week 8 (Reset Baseline) to Week 104 (with no 12-week confirmed EDSS progression determined at Week 116). NEDA was defined as follows: no EDSS progression (12-week sustained); no relapses; no Gd+ lesions; no new or enlarging T2 hyperintense lesions over 48 weeks after resetting the Baseline at Week 8 to remove contribution of CUA lesions that occurred prior to Week 8, when natalizumab was not yet active. The EDSS quantifies disability in 8 functional systems. The final EDSS score is an ordinal clinical rating scale ranging from 0 (normal neurologic examination) to 10 (death due to MS) in half-point increments.
Time Frame: from Week 8 (Reset Baseline) to Week 104
Population: as for outcome 1
Arm/Group | Natalizumab
Number analyzed (Participants) | 0

4. Secondary Outcome: Pre- and Post-Natalizumab Infusion Annualized Relapse Rate (ARR) Comparison at Month 12
Description: An MS relapse was defined as the onset of new or recurrent neurological symptoms lasting at least 24 hours, accompanied by new objective abnormalities on a neurological examination, and not explained solely by non-MS processes such as fever, infection, severe stress, or drug toxicity. 95% confidence interval is based on a Poisson regression model.
Time Frame: From 12 months prior to natalizumab infusion and 12 months post-natalizumab infusion
Population: Intent-to-treat population: participants who received at least 1 infusion of study treatment and had an assessment.
Measure: Number (95% Confidence Interval); unit: relapses per subject-year
Arm/Group | Natalizumab
Number analyzed (Participants) | 47
relapses per subject-year
  12 months pre-natalizumab infusion | 1.553 [1.306 to 1.847]
  12 months post-natalizumab infusion | 0.159 [0.076 to 0.331]

5. Secondary Outcome: Change in MSIS-29 Physical Impact Scores From Baseline (Day -1) to Reset Baseline (Week 8)
Description: The MSIS-29 is a brief self-administered MS-specific instrument measuring physical (20 items) and mental/psychological (9 items) impact of MS. The physical score is generated by summing individual items and then transforming to a scale with a range of 0 to 100, where high scores indicate worse health.
Time Frame: Baseline (Day -1) to Reset Baseline (Week 8)
Population: Intent-to-treat population: participants who received at least 1 infusion of study treatment and had an assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Natalizumab
Number analyzed (Participants) | 45
units on a scale | -2.53 (12.42)

ADVERSE EVENTS:
Time Frame: From Screening through end of study. Duration of study treatment was up to 13 months.
Description: SAEs only were collected per protocol. Events were not coded by MedDRA.
Arm/Group | Natalizumab
Serious Adverse Events (participants affected / at risk) | 2/47
Other Adverse Events (participants affected / at risk) | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Natalizumab (N=47)
Syncope (Nervous system disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
As a result of early study termination and limited available data, no meaningful conclusions can be drawn.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreement is subject to confidentiality but generally the PI can publish, for noncommercial purposes only, results and methods of the trial, but no other Sponsor Confidential Information. PI must give Sponsor no less than 60 days to review any manuscript for a proposed publication and must delay publication for up to an additional 90 days thereafter if Sponsor needs to file any patent application to protect any of Sponsor's intellectual property contained in the proposed publication.